CLINICAL TRIAL: NCT06214052
Title: A Phase 2a, Randomized, Double-Blind (Sponsor Unblinded), Placebo-Controlled, Study to Investigate the Antiviral Effect, Safety, Tolerability and Pharmacokinetics of VH4524184 in HIV-1 Infected Treatment Naïve Adults
Brief Title: VH4524184 Proof-of-Concept in Treatment-Naïve Adults Living With HIV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218806; 2023-507173-18-00 (Other: EU CT Number)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency virus; Proof of concept; Antiviral Agents; Virus Diseases
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Virus Diseases | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Data will be collected in a double-blind manner during the monotherapy phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- VH4524184 Dose 1 (Experimental): Participants received VH4524184, administered as Dose 1 (low dose) on Day 1, Day 4, and Day 7. On Day 10, participants began open-label standard-of-care (SOC) antiretroviral therapy (ART), which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
  Interventions: Drug: VH4524184; Drug: Antiretroviral therapy
- VH4524184 Dose 2 (Experimental): Participants received VH4524184, administered as Dose 2 (medium dose) on Day 1, Day 4, and Day 7. On Day 10, participants began open-label SOC ART, which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
  Interventions: Drug: VH4524184; Drug: Antiretroviral therapy
- VH4524184 Dose 3 (Experimental): Participants received VH4524184, administered as Dose 3 (high dose) on Day 1, Day 4, and Day 7. On Day 10, participants began open-label SOC ART, which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
  Interventions: Drug: VH4524184; Drug: Antiretroviral therapy
- Placebo (Placebo Comparator): Participants received matching Placebo to the study intervention on Day 1, Day 4, and Day 7. On Day 10, participants began open-label SOC ART, which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
  Interventions: Drug: Matching Placebo; Drug: Antiretroviral therapy

INTERVENTIONS:
Drug: VH4524184 — VH4524184 was administered as tablets orally at Day 1.
  Arms: VH4524184 Dose 1; VH4524184 Dose 2; VH4524184 Dose 3
Drug: Matching Placebo — VH4524184 Matching Placebo was administered as tablets orally at Day 1.
  Arms: Placebo
Drug: Antiretroviral therapy — Antiretroviral therapy was administered as available and as per investigator's recommendation.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, ability of VH4524184 when given alone to reduce the amount of HIV (viral load) in people with HIV-1 infection who have never received antiretroviral therapy (treatment-naïve). Data from this study will be used to decide how VH4524184 can be best included in a full-treatment regimen for HIV-1 in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive at the time of signing the informed consent.
* Participants who are overtly healthy (other than HIV infection) as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Positive HIV antibody test
* Documented HIV infection and Screening plasma HIV-1 RNA ≥ 3,000 copies/mL. A single repeat of this test is allowed within a single Screening period to determine eligibility.
* Screening CD4+ T-cell count ≥200 cells/mm3
* Treatment-naïve: No antiretrovirals (ARVs, in combination or monotherapy) received after the diagnosis of HIV-1 infection.
* HIV Pre-exposure or post-exposure prophylaxis: No prior use of any INSTI (including cabotegravir) for HIV pre-exposure or post-exposure prophylaxis.
* Body weight ≥50.0 kg (110 lbs.) for men and ≥45.0 kg (99 lbs) for women and BMI within the range 18.5-31.0 kg/m2 (inclusive - applies to males and females).
* A participant of childbearing potential must have a negative serum hCG test at screening, and negative urine hCG test at Day 1, before the first dose of study intervention.
* If a urine test cannot be confirmed as negative (e.g. ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease risk for inclusion of a female with an early undetected pregnancy.
* Capable of giving signed informed consent
* Participant must be willing and able to start standard-of-care ART as selected with the investigator on Study Day 10.

Exclusion Criteria:

* Participants with primary HIV infection. Any evidence of an active CDC Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy during the study. Untreated syphilis infection [positive RPR at screen] without documentation of treatment. Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; or other localized malignancies
* Any pre-existing physical or mental condition which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Any history of significant underlying psychiatric disorder, or a clinical assessment of suicidality based on the responses on the eCSSRS.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders, that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome or sudden cardiac death. Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of study drug administration.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing. Specific medications listed in Section 6.9.1 may be allowed.
* Participants who require concomitant medications known to be associated with a prolonged QTc.
* Participants receiving any protocol-prohibited medication(s) and who are unwilling or unable to switch to an alternate medication).
* The participant has ever received an investigational HIV vaccine (immunotherapeutic or immunomodulatory).
* Exposure to an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study intervention.
* Participation in the study would result in donation of blood in excess of 500 mL within 56 days.
* Exposure to more than four new investigational drugs or vaccines within 12 months prior to the first dosing day.
* Current enrollment or past participation within the last 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.

Diagnostic Assessments

* Presence of HBsAg or HBcAb at screening
* Positive Hepatitis C antibody test result at Screening
* Positive Hepatitis C RNA test result at Screening.
* Creatinine clearance (eGFR) of < 60 mL/min/1.73 m2 using CKD-EPI equation (2021).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (5):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, West Hollywood, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Orlando, Florida
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
- Canada (2):
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Milan, Italy
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 2 of the study was optional and was not selected for enrollment following interim analysis of part 1 based on Pharmacokinetic/Pharmacodynamic modelling and preliminary clinical data.
Period: Monotherapy Period (Day 1 to Day 10)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Started | 6 | 6 | 7 | 3
Completed | 6 | 6 | 7 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Follow-Up Period(Day 11 to Day 38)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Started | 6 | 6 | 7 | 3
Completed | 6 | 6 | 7 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 22
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 34.2 (10.61) | 36.7 (16.18) | 33.9 (12.52) | 29.3 (3.79) | 34.1 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 3
  Male | 6 | 4 | 6 | 3 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The "All Other Races" category, which includes american indian or alaska native, asian, black or african american, and white (where 0 < n < 11), represents the combination of these race categories into a single category to ensure participant confidentiality and privacy.
  Participants
    All Other Races | 6 | 6 | 7 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Monotherapy: Maximum Change From Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA)
Description: Plasma samples were collected for the quantitative analysis of plasma HIV-1 RNA. The maximum change from baseline was calculated by determining the largest change from baseline value across all assessment timepoints during the monotherapy period. This is identified by subtracting the lowest post-dose visit value up to Day 10 (inclusive) from the baseline value. The baseline was defined as the most recent pre-dose assessment with a valid, non-missing value, including measurements from any unscheduled visits.
Time Frame: At Day 10
Population: Analysis was performed on Full Analysis Set (FAS), which included all randomized participants who received at least 1 full dose of study intervention.
Measure: Mean (Standard Deviation); unit: Copies per milliliter (copies/mL)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Copies per milliliter (copies/mL) | -1.17 (0.460) | -2.15 (0.254) | -2.31 (0.463) | -0.28 (0.370)

2. Secondary Outcome: Monotherapy and Follow-up: Number of Participants With Any Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE can be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Any AEs = occurrence of the symptom regardless of intensity grade.
Time Frame: Day 1 to Day 38
Population: Analysis was performed on the Safety Set, which included all randomized participants who received at least one partial or full dose of the study intervention. As pre-specified in the protocol, the outcome measure data are reported for monotherapy and FU periods combined that includes all participants and all doses administered during the specified duration. Each participant is counted once across both the periods, reflecting the total number of participants affected by any adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Participants | 4 | 6 | 5 | 2

3. Secondary Outcome: Monotherapy and Follow-up: Number of Participants With AEs by Severity
Description: The severity was assessed using The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) Version 2.1 where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening and Grade 5 = Death.
Time Frame: Day 1 to Day 38
Population: Analysis was performed on Safety Set. As pre-specified in the protocol, the outcome measure data are reported for monotherapy and FU periods combined that includes all participants and all doses administered during the specified duration. Each participant is counted once across both the periods, reflecting the total number of participants affected by any adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Participants
  Grade 1 | 3 | 4 | 3 | 1
  Grade 2 | 1 | 2 | 2 | 1
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

4. Secondary Outcome: Monotherapy: Number of Participants With AEs Leading to Study Treatment Discontinuation
Time Frame: Day 1 to Day 7
Population: Analysis was performed on Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Monotherapy and Follow-up: Change From Baseline for Liver Panel Laboratory Parameters: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP)
Description: Blood samples were collected at the indicated timepoints.
Time Frame: At Baseline (Day 1), Day 2, Day 4, Day 7, Day 10, Day 17, Day 24, Day 31 and Day 38
Population: Analysis was performed on Safety Set. As pre-specified in the protocol, the outcome measure data are reported for monotherapy and FU periods combined that includes all participants and all doses administered during the specified timepoints.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
International units per liter (IU/L)
  ALT, Baseline (Day 1) | 25.5 (15.35) | 26.0 (9.27) | 30.4 (20.82) | 21.0 (7.21)
  ALT, Day 2 | 0.0 (4.20) | 1.3 (2.50) | 4.3 (11.70) | 0.0 (4.00)
  ALT, Day 4 | 2.2 (4.54) | 0.5 (4.42) | 0.0 (12.41) | -1.0 (1.00)
  ALT, Day 7 | 0.2 (3.25) | -3.5 (5.36) | -6.4 (14.39) | -1.3 (5.86)
  ALT, Day 10 | 4.5 (5.79) | -5.5 (5.82) | -6.1 (16.95) | 8.3 (16.50)
  ALT, Day 17: number analyzed (Participants) | 6 | 5 | 7 | 3
  ALT, Day 17 | 6.7 (15.10) | -7.0 (6.24) | -8.0 (13.99) | -3.0 (8.72)
  ALT, Day 24 | -1.7 (6.15) | 1.2 (12.22) | -8.6 (14.41) | -4.3 (4.51)
  ALT, Day 31: number analyzed (Participants) | 5 | 6 | 7 | 3
  ALT, Day 31 | -2.8 (10.31) | 0.2 (7.31) | -10.4 (11.84) | -5.0 (4.58)
  ALT, Day 38 | -2.8 (8.26) | -2.5 (9.16) | -13.0 (16.67) | -3.0 (5.57)
  AST, Baseline (Day 1) | 29.7 (24.64) | 26.5 (11.45) | 25.9 (8.76) | 22.3 (11.68)
  AST, Day 2 | -1.3 (6.65) | -1.2 (4.96) | 2.6 (10.06) | 0.0 (3.46)
  AST, Day 4 | 2.2 (3.06) | -3.2 (9.02) | -2.9 (6.12) | 1.3 (3.06)
  AST, Day 7 | -0.3 (3.67) | -4.8 (6.97) | -4.9 (6.57) | -0.7 (4.73)
  AST, Day 10 | 9.7 (17.82) | -6.2 (8.47) | -4.7 (7.45) | 2.0 (11.79)
  AST, Day 17: number analyzed (Participants) | 6 | 5 | 7 | 3
  AST, Day 17 | 22.0 (47.41) | -9.0 (5.83) | -5.1 (7.36) | -1.3 (8.74)
  AST, Day 24 | 1.2 (8.01) | -4.3 (6.59) | -3.3 (6.73) | -4.0 (7.00)
  AST, Day 31: number analyzed (Participants) | 5 | 6 | 7 | 3
  AST, Day 31 | -0.8 (6.30) | -3.0 (4.20) | -2.4 (6.45) | -3.0 (5.20)
  AST, Day 38 | -4.7 (14.05) | -4.7 (5.54) | -6.0 (9.36) | 0.3 (8.02)
  ALP, Baseline (Day 1) | 81.3 (32.51) | 70.3 (15.76) | 72.9 (10.06) | 103.7 (56.00)
  ALP, Day 2 | 3.3 (9.14) | 2.5 (6.69) | 0.6 (3.26) | 7.3 (13.58)
  ALP, Day 4 | 2.5 (9.18) | -0.2 (3.13) | 2.9 (5.84) | 13.3 (18.01)
  ALP, Day 7 | 3.7 (6.50) | -4.0 (3.63) | -2.6 (4.72) | 2.7 (15.82)
  ALP, Day 10 | 4.2 (3.92) | -1.7 (6.53) | 2.1 (3.89) | 5.7 (13.65)
  ALP, Day 17: number analyzed (Participants) | 6 | 5 | 7 | 3
  ALP, Day 17 | 4.5 (5.09) | 0.0 (3.74) | 0.9 (6.72) | 8.3 (4.93)
  ALP, Day 24 | 3.2 (2.86) | -0.2 (5.19) | -0.7 (6.80) | -1.3 (17.01)
  ALP, Day 31: number analyzed (Participants) | 5 | 6 | 7 | 3
  ALP, Day 31 | 5.2 (3.90) | 0.3 (12.60) | 0.1 (9.01) | 20.3 (14.36)
  ALP, Day 38 | 4.5 (3.51) | 0.2 (14.33) | -0.6 (5.83) | -3.0 (21.17)

6. Secondary Outcome: Monotherapy and Follow-up: Change From Baseline for Liver Panel Laboratory Parameter: Bilirubin
Description: Blood samples were collected at the indicated timepoints.
Time Frame: At Baseline (Day 1), Day 2, Day 4, Day 7, Day 10, Day 17, Day 24, Day 31 and Day 38
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Micromoles per liter (μmol/L)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Micromoles per liter (μmol/L)
  Baseline (Day 1) | 8.2935 (5.93914) | 5.6145 (3.21992) | 5.9117 (3.21410) | 8.0370 (5.75333)
  Day 2 | 1.0545 (3.03093) | 0.2565 (1.32787) | 1.1481 (1.75421) | -0.7410 (4.86174)
  Day 4 | 1.4820 (5.38437) | 0.8550 (2.93204) | 1.6856 (3.71694) | -3.2490 (5.08132)
  Day 7 | -1.5105 (4.25706) | 2.1660 (2.20230) | -0.8306 (2.63700) | -1.8813 (5.60653)
  Day 10 | 2.2515 (6.11541) | 0.7695 (3.53892) | 0.3176 (2.28020) | -3.0210 (3.16389)
  Day 17: number analyzed (Participants) | 6 | 5 | 7 | 3
  Day 17 | 0.7980 (7.47774) | 0.1368 (3.23863) | 0.4641 (3.39097) | 1.7670 (4.44052)
  Day 24 | 1.7100 (6.10927) | 0.2280 (3.65583) | 1.3436 (3.54789) | -0.5130 (2.68748)
  Day 31: number analyzed (Participants) | 5 | 6 | 7 | 3
  Day 31 | -0.2052 (7.41576) | 0.0285 (1.40768) | 0.3909 (2.62828) | 0.8550 (4.42292)
  Day 38 | 1.7100 (5.46665) | -0.1712 (3.59512) | 0.2931 (1.14163) | -3.1923 (3.60425)

7. Secondary Outcome: Monotherapy and Follow-up: Change From Baseline for Liver Panel Laboratory Parameter: Protein
Description: Blood samples were collected at the indicated timepoints.
Time Frame: At Baseline (Day 1), Day 2, Day 4, Day 7, Day 10, Day 17, Day 24, Day 31 and Day 38
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Grams per liter
  Baseline (Day 1) | 76.5 (4.55) | 75.5 (3.39) | 77.1 (5.49) | 70.0 (5.57)
  Day 2 | 2.8 (3.60) | 2.2 (3.31) | 0.7 (3.30) | 5.7 (1.53)
  Day 4 | 4.3 (4.37) | 1.5 (2.66) | 2.1 (2.97) | 2.0 (1.00)
  Day 7 | 2.0 (3.63) | -1.3 (2.34) | -1.9 (3.89) | -1.0 (1.00)
  Day 10 | 2.2 (2.40) | -0.7 (3.14) | 1.6 (2.64) | 0.3 (2.08)
  Day 17: number analyzed (Participants) | 6 | 5 | 7 | 3
  Day 17 | 1.2 (3.25) | 0.4 (2.30) | 0.1 (5.21) | 7.3 (4.16)
  Day 24 | 0.8 (3.06) | 0.3 (4.46) | 0.6 (4.43) | 2.0 (3.00)
  Day 31: number analyzed (Participants) | 5 | 6 | 7 | 3
  Day 31 | 0.4 (4.56) | -0.2 (5.23) | -0.9 (3.80) | 8.3 (4.51)
  Day 38 | 0.5 (2.26) | -1.3 (4.68) | -1.4 (4.35) | 2.0 (4.58)

8. Secondary Outcome: Monotherapy and Follow-up: Number of Participants With Maximum Toxicity Grade Increase Relative to Baseline in Liver Panel Laboratory Parameters: ALT, AST, ALP, Bilirubin
Description: Liver panel parameters assessed were: ALT, AST, ALP, bilirubin. The parameters were graded according to DAIDS grading table Version 2.1 where grades were defined based on numeric criteria as follows Grade 0: participants with missing baseline values; Grade 1: Mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. An increase is defined as an increase in grade relative to baseline grade.
Time Frame: From Baseline (Day 1) and up to Day 38
Population: Analysis was performed on Safety Set. As pre-specified in the protocol, the outcome measure data are reported for monotherapy and FU periods combined that includes all participants and all doses administered during the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Participants
  ALT, Increase to Grade 1 | 0 | 1 | 1 | 0
  ALT, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 0 | 0 | 1 | 0
  AST, Increase to Grade 2 | 1 | 0 | 0 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 1 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0
  Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0

9. Secondary Outcome: Monotherapy and Follow-up: Number of Participants With Maximum Toxicity Grade Increase Relative to Baseline in Liver Panel Laboratory Parameters: Protein
Description: Participants are categorized based on changes in their liver panel laboratory parameters (protein) to 'Low,' 'Normal,' or 'High,' unless there is no change in their initial category. Participants whose lab values remain unchanged (e.g., 'High' to 'High') or whose values return to normal are recorded in the 'To Normal or No Change' category. Participants may be counted in both the 'To Low' and 'To High' categories if their values fluctuate between these states. As a result, the percentages may exceed 100% due to dual categorization. Participants with a missing baseline value are assumed to have a normal baseline value.
Time Frame: From Baseline (Day 1) and up to Day 38
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
Participants
  To Low | 0 | 0 | 0 | 0
  To Normal or No Change | 4 | 4 | 5 | 2
  To High | 2 | 2 | 2 | 1

10. Secondary Outcome: Monotherapy: Maximum Observed Plasma Drug Concentration (Cmax) of VH4524184
Description: Blood samples were collected at indicated time points for Pharmacokinetic (PK) analysis of VH4524184.
Time Frame: At Day 1 and Day 7
Population: Analysis was performed on PK Set, which included All participants in the Safety analysis set who had at least 1 non-missing PK assessment. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3
Number analyzed (Participants) | 6 | 6 | 7
Nanogram per milliliter (ng/mL)
  Day 1 | 1332.57 (16.78) | 6173.61 (30.71) | 23589.70 (32.39)
  Day 7 | 1488.59 (32.06) | 7112.60 (16.59) | 23069.92 (45.77)

11. Secondary Outcome: Monotherapy: Time to Maximum Observed Plasma Drug Concentration (Tmax) of VH4524184
Description: Blood samples were collected at indicated time points for PK analysis of VH4524184.
Time Frame: At Day 1 and Day 7
Population: Analysis was performed on PK Set. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3
Number analyzed (Participants) | 6 | 6 | 7
hours
  Day 1 | 3.13 [1.0 to 5.0] | 4.00 [2.0 to 5.0] | 2.00 [1.0 to 5.0]
  Day 7 | 4.00 [0.5 to 5.1] | 4.49 [1.0 to 6.0] | 2.13 [1.0 to 4.0]

12. Secondary Outcome: Monotherapy: Plasma Concentration of VH4524184 at Day 10
Description: Blood samples was collected at indicated time point for PK analysis of VH4524184.
Time Frame: At Day 10
Population: Analysis was performed on PK Set. Only participants with data available at the specified timepoint were included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3
Number analyzed (Participants) | 6 | 6 | 7
ng/mL | 127.5 (75.59) | 523.5 (324.50) | 1328.3 (486.99)

13. Secondary Outcome: Monotherapy: Correlation of VH4524184 Cmax With Maximum Plasma HIV-1 RNA Log 10 Change From Baseline Through Day 10
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value was the latest pre-dose assessment with a non-missing value. Change from baseline is defined as post-dose visit value minus baseline value. Statistical analysis for relationship between PK parameter (Cmax) and PD measure (change from baseline in logarithm to base 10 (log10) values for maximum plasma HIV-1 RNA) were explored using an Emax non-linear mixed-effects model. The model parameters estimated were maximum response (Emax) which is defined as the maximum change (at infinite exposure) and EC50 which defines the PK parameter value that attains 50 percent (%) of the maximal effect
Time Frame: From Day 1 to Day 10
Population: Analysis was performed on PK Set. Only participants with data available at the specified duration were included in this analysis.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3
Number analyzed (Participants) | 6 | 6 | 7
Log10 copies/mL | -1.17 (0.460) | -2.15 (0.254) | -2.31 (0.463)
Statistical Analysis 1: Comparison: VH4524184 Dose 1 vs VH4524184 Dose 2 vs VH4524184 Dose 3; Test type: Other; Emax = -2.69, Standard Error of Mean 5
Statistical Analysis 2: Comparison: VH4524184 Dose 1 vs VH4524184 Dose 2 vs VH4524184 Dose 3; Test type: Other; EC50 = 1.88, Standard Error of Mean 26

14. Secondary Outcome: Monotherapy: Number of Participants With Treatment-emergent Genotypic Resistance
Description: Plasma samples were collected to assess treatment emergent Genotypic Resistance.
Time Frame: At Baseline (Day 1) and Day 10
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Day 1 | 0 | 0 | 0
  Day 10 | 0 | 0 | 0

15. Secondary Outcome: Monotherapy: Number of Participants With Treatment-emergent Phenotypic Resistance
Description: Plasma samples were collected to assess treatment emergent Phenotypic Resistance.
Time Frame: At Baseline (Day 1) and Day 10
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Day 1 | 0 | 0 | 0
  Day 10 | 0 | 0 | 0

16. Secondary Outcome: Monotherapy: Change From Baseline in Cluster of Differentiation 4 (CD4+) T-cell Counts at Day 10
Description: Blood samples were collected for assessment of T-cells subsets (CD4+ T-cells count) by flow cytometry at Day 10 compared to Baseline.
Time Frame: At Day 10 compared to Baseline (Day 1)
Population: Analysis was performed on Safety Set. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Mean (Standard Deviation); unit: CD4+ million cells per Liter (10^6/L)
Arm/Group | VH4524184 Dose 1 | VH4524184 Dose 2 | VH4524184 Dose 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 3
CD4+ million cells per Liter (10^6/L) | 131.333 (98.4473) | 68.667 (122.1191) | 47.000 (45.9093) | 63.667 (216.1512)

ADVERSE EVENTS:
Time Frame: Serious AEs (SAEs) and Non-serious AEs were assessed from Day 1 until the final visit in the Follow-up Period (at Day 38)
Description: Adverse events are reported individually for the Monotherapy and Follow-Up period from the Safety Set. Participants are counted in each period based on the occurrence and frequency of events.
Groups:
- VH4524184 Dose 1_Monotherapy: Participants received VH4524184 Dose 1 (low dose) on Day 1, Day 4, and Day 7.
- VH4524184 Dose 2_Monotherapy: Participants received VH4524184 Dose 2 (medium dose) on Day 1, Day 4, and Day 7.
- VH4524184 Dose 3_Monotherapy: Participants received VH4524184 Dose 3 (high) on Day 1, Day 4, and Day 7.
- Placebo_Monotherapy: Participants received matching Placebo to the study intervention on Day 1, Day 4, and Day 7.
- VH4524184 Dose 1_Follow-up: Participants received VH4524184, administered as Dose 1 (low dose) on Day 1, Day 4, and Day 7. On Day 10, participants began open-label standard-of-care (SOC) antiretroviral therapy (ART), which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
- VH4524184 Dose 2_Follow-up: Participants received VH4524184, administered as Dose 2 (medium dose) on Day 1, Day 4, and Day 7. On Day 10, participants began open-label SOC ART, which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
- VH4524184 Dose 3_Follow-up: Participants received VH4524184, administered as Dose 3 (high dose) on Day 1, Day 4, and Day 7. On Day 10, participants began open-label SOC ART, which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
- Placebo_Follow-up: Participants received matching Placebo to the study intervention on Day 1, Day 4, and Day 7. On Day 10, participants began open-label SOC ART, which was selected by the investigator and locally sourced. Participants were monitored weekly until Day 38.
Arm/Group | VH4524184 Dose 1_Monotherapy | VH4524184 Dose 2_Monotherapy | VH4524184 Dose 3_Monotherapy | Placebo_Monotherapy | VH4524184 Dose 1_Follow-up | VH4524184 Dose 2_Follow-up | VH4524184 Dose 3_Follow-up | Placebo_Follow-up
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/3 | 0/6 | 0/6 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/3 | 0/6 | 0/6 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 3/7 | 2/3 | 4/6 | 5/6 | 4/7 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VH4524184 Dose 1_Monotherapy (N=6) | VH4524184 Dose 2_Monotherapy (N=6) | VH4524184 Dose 3_Monotherapy (N=7) | Placebo_Monotherapy (N=3) | VH4524184 Dose 1_Follow-up (N=6) | VH4524184 Dose 2_Follow-up (N=6) | VH4524184 Dose 3_Follow-up (N=7) | Placebo_Follow-up (N=3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT06214052/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT06214052/SAP_001.pdf